CLINICAL TRIAL: NCT05113485
Title: A Fiber-diverse, Anti-inflammatory Diet and Aerobic Exercise Reduce Risk of Breast Cancer Recurrence
Brief Title: UCLA Breast Cancer Survivor Health Promotion Research Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, William J. McCarthy, Ph.D., Adjunct Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B27IB3856
Record Dates: First submitted 2021-10-19; First posted 2021-11-09 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
Keywords: obesity; physical activity; fiber diversity; calorie restriction; inflammation
MeSH Terms: conditions — Breast Neoplasms; Obesity; Motor Activity; Inflammation | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The two lifestyle change interventions feature a similar exercise prescription and the same sequence of intervention contacts (2 virtual home visits; 2 virtual group education sessions, 7 individual telephone coaching sessions) but differ in dietary approach. The DPP-based diet approach prescribes desired weight loss in overweight breast cancer survivors by restricting daily calorie intake and promoting increased calorie expenditure via physical activity. The HMAFs approach prescribes consuming an optimal six microbiota-accessible foods unaccompanied by pro-inflammatory food components such as saturated fat or added sugar as well as engaging regularly in exercise that elevates the heart rate and reduces inflammation. Only 20 percent of daily calories need to be devoted to HMAFs; the remaining calories can come from daily food choices conforming to the 2020-2025 Dietary Guidelines for Americans.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All assessments will be conducted by project personnel blind to the study participants' randomization status. The investigators responsible for helping participants complete the Automated Self-administered 24-hour (ASA 24) dietary recalls and for assessing their body composition via dual x-ray absorptiometry (DXA) will be kept blind to the study participants' randomization status. Investigators will be kept blind to participant assignment to condition by having the two health coaches refer to their patients by an arbitrary, unique study identifier during weekly debriefings when the study progress by individual participants might be discussed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Prevention Program-based lifestyle change intervention (DPP) (Active Comparator): The Diabetes Prevention Program-based lifestyle change intervention (DPP) is designed to help overweight breast cancer survivors to reduce their risk of breast cancer recurrence by reducing their excess body fat.
  Interventions: Behavioral: Diabetes Prevention Program-based lifestyle change intervention (DPP)
- Highly Microbiota-Accessible Foods (HMAFs) intervention (Experimental): The Highly Microbiota-Accessible Foods (HMAFs) lifestyle change intervention is designed to help overweight breast cancer survivors reduce their risk of breast cancer recurrence by reducing their elevated low-grade inflammation.
  Interventions: Behavioral: Highly Microbiota-Accessible Foods (HMAFs) intervention

INTERVENTIONS:
Behavioral: Diabetes Prevention Program-based lifestyle change intervention (DPP) — The DPP condition consists of 11 health education sessions over 12 weeks, including 2 virtual home visits, two virtual group education sessions and 7 telephone coaching calls. These sessions will teach DPP-based lessons on how to lose excess body fat through calorie restriction and increased physical activity. All dietary and physical activity recommendations are intended to be consistent with federal nutrition and physical activity guidelines.
  Arms: Diabetes Prevention Program-based lifestyle change intervention (DPP)
Behavioral: Highly Microbiota-Accessible Foods (HMAFs) intervention — The Highly Microbiota-Accessible Foods (HMAFs) intervention approach includes 11 health education sessions, including two virtual home visits, two virtual group education sessions, and 7 telephone coaching sessions. These sessions are designed to help study participants to identify and consume optimally 6 daily instances of minimally processed, fiber-rich food sources, drawn from all four of the MyPlate.gov categories: vegetables, fruits, whole grains and plant-based protein-rich foods (e.g., legumes, nuts and seeds). Increased physical activity is also recommended as a way to optimize the microbial conversion of fiber-rich food sources to short chain fatty acids, which are then expected to reduce excess low-grade inflammation.
  Arms: Highly Microbiota-Accessible Foods (HMAFs) intervention

SUMMARY:
Pilot randomized controlled parallel group behavior change comparative effectiveness trial involves 30 breast cancer survivors interested in losing excess body fat. Both interventions include dietary + exercise prescriptions that hold promise for reducing the survivors' risk of cancer recurrence. Both interventions are consistent with the Dietary Guidelines for Americans but the Diabetes Prevention Program (DPP)-based approach focuses on weight loss through calorie restriction and increased physical activity while the Highly Microbiota-Accessible Foods (HMAFs) approach is intended to be a low-numeracy version of a Mediterranean-style diet and increased physical activity. The DPP approach is considered to be a high-numeracy intervention because it requires that consumers keep track of all calories consumed and expended per day and to endeavor to maintain a calorie deficit each day during the active weight loss phase. For both conditions, the 12 to 13-week intervention includes 2 virtual home visits, 2 virtual group education sessions and 7 telephone or Zoom-based coaching sessions by well-trained intervenors. Assessments occur at baseline and six months, with systemic inflammation (high sensitivity C-reactive protein) being the primary outcome measure and visceral fat being a secondary outcome. Other prespecified secondary outcomes include gut microbiota alpha-1 diversity, insulin resistance, HDL-cholesterol, daily count of highly microbiota-accessible foods, waist circumference, BMI, systolic blood pressure, ratio of fecal Proteobacteria to short chain fatty acid-generating bacteria and health-related quality of life.

DETAILED DESCRIPTION:
Background. The human gut microbiota influences obesity status and inflammation, two major risk factors for postmenopausal breast cancer recurrence. Whether an exercise and dietary intervention designed to optimize gut microbiota composition might reduce risk for breast cancer recurrence is unknown. To improve the gut microbiota composition, the investigators propose teaching postmenopausal breast cancer survivors to allocate about 20% of their daily calorie intake to consuming a daily count of six fiber-rich, minimally processed, plant-based food choices that comply with federal MyPlate.gov diet recommendations. Preliminary data suggest that the investigators' Highly-Microbiota-Accessible Foods (HMAFs) approach will yield cardiometabolic outcomes equal to or better than those achieved by the traditional Diabetes Prevention Program (DPP) calorie restriction approach at 6 months follow-up. Because breast cancer recurrence risk covaries with cardiometabolic risks, the lower cardiometabolic risk of the HMAFs approach should be associated with reduced risk of breast cancer recurrence.

Hypotheses. The greater diversity of fiber-rich, minimally processed plant foods consumed in the HMAFs condition relative to the DPP condition will result in greater changes in HMAFs participants compared to DPP participants from baseline to 6 months follow-up in the following measures: (primary hypothesis) reduce high sensitivity C-reactive protein, (secondary hypotheses) reduce visceral body fat and increase alpha-1 diversity of gut microbes and increase health-related quality of life.

To test these hypotheses, the research objectives include the following specific aims: 1) Recruit a diverse sample of 30 overweight or obese postmenopausal survivors with stage I, II and IIIa breast cancer; randomly allocate them to two lifestyle change intervention conditions, 2) Obtain baseline and 6-month follow-up assessments of: low grade systemic inflammation, body composition including visceral fat estimation, cardiorespiratory fitness, inflammatory and cardiometabolic biomarkers, fecal samples, and quality of life, 3) Conduct two parallel, three-month behavior change interventions, contrasting the 6-count HMAFs approach with the traditional DPP calorie restriction approach , and 4) Use results to design a ramped-up randomized factorial trial.

If hypotheses are confirmed, the low-numeracy HMAFs approach may, for low-income survivors, be a practical alternative to traditional high-numeracy calorie restriction approaches to reducing risk of breast cancer recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. At least 6 months since breast cancer diagnosis and up to 4 years since diagnosis.
2. Between 50 and 75 years of age.
3. Diagnosed with localized steroid hormone receptor-positive breast cancer, up to stage IIIa.
4. At least 6 months post chemotherapy or radiation treatment.
5. Subjects must be in good health as determined by medical history, physical examination, and clinical laboratory measurements.
6. No broad-spectrum antibiotic use in the last two months.
7. Body mass index between 27 and 38 based on self-reported height and weight and between 25 and 40 based on objective assessment of height and weight.
8. Willing to complete assessments at baseline, 3 months and 6 months follow-up

Exclusion Criteria:

1. Diagnosed with metastatic breast cancer
2. Currently undergoing chemotherapy or radiation treatment
3. Immunoglobulin-E (IgE)-mediated food allergies, or any medical condition requiring mandatory dietary restrictions
4. Significant cardiac, pulmonary, renal, liver or psychiatric disease.
5. Muscular, orthopedic, or cardiovascular limitations that would prevent full participation in exercise

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
High-sensitivity C-Reactive Protein (CRP) | Change from baseline to 6 months follow-up
  CRP is commonly used by researchers as a biomarker for systemic inflammation.

SECONDARY OUTCOMES:
Visceral fat as assessed by DXA | Change from baseline to six months follow-up
  Visceral fat is also known as intra-abdominal fat. It is located inside the peritoneal cavity, packed in between internal organs and torso. It is the most metabolically active adipose tissue and positively associated with systemic inflammation.
Shannon index of alpha diversity of fecal microbial species | Change from baseline to six months follow-up
  Fecal DNA from the V4 region of the 16S ribosomal RNA will be amplified, sequenced and filtered for quality before statistical analysis. The Shannon index measures both gene richness and evenness.
Number of highly microbiota-accessible foods consumed per day | Change from baseline to six months follow-up
  From participants' 24-hour diet recalls - The daily sum of different carbohydrate-rich food sources minimally processed and unaccompanied by pro-inflammatory components, especially saturated fat and added sugar.

OTHER OUTCOMES:
Insulin resistance | Change from baseline to six months follow-up
  Homeostatic Model Assessment-Insulin Resistance (HOMA-IR) is a recognized measure of insulin resistance, calculated from fasting glucose and fasting insulin values
Waist circumference | Change from baseline to six months follow-up
  Waist circumference is measured via non-stretchable measuring tape around the waist at a midpoint between the lowest rib and the iliac crest, upon breath exhalation.
Body mass index (BMI) | Change from baseline to six months follow-up
  Height measured via wall-mounted stadiometer and weight measured via calibrated digital scale will be used to compute BMI ((kg/(m x m))
Systolic blood pressure (mm) | Change from baseline to six months follow-up
  Regularly calibrated digital sphygmomanometer will be used to assess the participant's resting systolic blood pressure in millimeters of mercury
Ratio of abundance of fecal Proteobacteria to fecal short chain fatty acid-generating bacteria | Change from baseline to six months follow-up
  Fecal DNA from the V4 region of the 16S ribosomal RNA will be amplified, sequenced and filtered for quality before statistical analysis. The ratio of fecal Proteobacterial abundance to the abundance of short-chain fatty acid-generating fecal microbes is expected to be reduced in healthier guts.
Health-related quality of life | Change from baseline to six months follow-up
  RAND Short Form-20 (SF-20) is recognized instrument for assessing participants' health-related quality of life. Minimum score = 0; maximum score = 100. Higher scores represent higher quality of life.
HDL-cholesterol | Change from baseline to six months follow-up
  Fasting serum HDL-cholesterol concentration expected to reflect the experimental differences in dietary patterns. Serum triglycerides will be generated as part of a standard lipid panel.

CONTACTS AND LOCATIONS:
Overall Officials: William J. McCarthy, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Cancer Prevention & Control Research, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be posted on the website of the UCLA Fielding School of Public Health for access by students and other investigators. Primary and secondary outcomes and demographic characteristics will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available 1 year after the completion of the final report.
Access Criteria: Bona fide researchers as determined by the University of California-Los Angeles (UCLA) Institutional Review Board (IRB) will be eligible to use the data.